CLINICAL TRIAL: NCT00388635
Title: A National, Multi-Center, Open-Label Study of Velcade in Combination With Melphalan and Prednisone (V-MP) in Older Untreated Multiple Myeloma Patients.
Brief Title: Velcade-Melphalan-Prednisone in Older Untreated Multiple Myeloma Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PET-VEL-2004-01
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Patients over 65 years old
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone

INTERVENTIONS:
Drug: Velcade — Phase I: Velcade, 1.0mg/m2-1.3mg/m2 in escalating doses every 6 weeks for 4 cycles Pase II: Velcade at optimal doses, twice a week (days 1, 4, 8, 11, 22, 25, 28 and 32) follow a rest period for 10 days (days 33 to 42)
Drug: Melphalan — Melfalán 9mg/m2 days 1 to 4, V.O, follow by a rest period of 38 days in phse I and II
Drug: Prednisone — Prednisone 60mg/m2 v.o days 1 to 4 follows by a rest period of 38 days (phase I and II)

SUMMARY:
This protocol is planned as a multicentric, national, open-label trial designed to evaluate, first, optimal dose of Velcade® (Bortezomib) in combination with melphalan and prednisone. After optimal dose is known, the second aim is evaluate safety and tolerance of V-MP plan, in respond terms, in a cohort of 60 patients. Finally, the entire results will be compared with those obtained from a series of 100 patients, all of them over 70 years old, diagnosed of Multiple Myeloma belonging to the GEM protocol finished in May 2003

DETAILED DESCRIPTION:
Multiple Myeloma is a neoplastic disorder of the last maturation stage of B cell, called plasmatic cell. It represents the second most common haematological neoplasia, after Non Hodgkin Lymphoma. The annual incidence is over 4 cases per 100.000. Multiple Myeloma is an invariably mortal disease. When illness advances, the reduction of infections resistance, the intense bones destruction (with bone pain, pathological fractures and hypercalcemia), anaemia, renal failure and, in a less frequency, neurological complications and hyperviscosity provoke severe morbidity and mortality. Five-year survival rate in patients with Multiple Myeloma treated with conventional chemotherapy is 29%. There is an urgent need of new therapeutic agents for the treatment of this disease

ELIGIBILITY:
Inclusion Criteria:

* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Age over 65 years.
* Patient recently diagnosed with symptomatic Multiple Myeloma based on standard criteria and that has not received any previous chemotherapy treatment for Multiple Myeloma.
* Patient has measurable disease, defined as follows:

For secretory multiple myeloma, measurable disease is defined as any quantifiable serum monoclonal protein value and, where applicable, urine light-chain excretion of ≥ 200 mg/24 hours.

For oligo or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan). In patients with oligo-secretory multiple myeloma, the serum and/or urine M-protein measurements are very low and difficult to follow for response assessment. In patients with non-secretory multiple myeloma, there is no M-protein in serum or urine.

* Patient has a Karnofsky performance status higher 60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline visit (Day 1 of Cycle 1, before study drug administration:

Platelet count ≥ 100x109/L, hemoglobin ≥ 8 g/dl and absolute neutrophil count (ANC) ≥ 1.0x109/L.

Corrected serum calcium < 14mg/dl. Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal. Alanine transaminase (ALT): ): ≤ 2.5 x the upper limit of normal. Total bilirubin: ≤1.5 x the upper limit of normal. Serum creatinine value ≤ 2mg/dl.

Exclusion Criteria:

* Patient previously received treatment with Velcade.
* Patient previously received treatment for Multiple Myeloma.
* Patient had major surgery within 4 weeks before enrollment.
* Patient has a platelet count < 100 x 109/L within 14 days before enrollment.
* Patient has an absolute neutrophil count < 1.0 x 109/L within 14 days before.
* Patient has < Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Patient has received other investigational drugs within 14 days before enrollment.
* Patient is known to be seropositive for the human immunodeficiency virus (HIV), Hepatitis B surface antigen-positive or active hepatitis C infection.
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.

Patient is enrolled in another clinical research study and/or is receiving an investigational agent for any reason.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-04; Primary Completion 2007-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determinate the efficacy of combination velcade, melphalan, prednisone | 1 year

SECONDARY OUTCOMES:
Assess safety and tolerability | 1 year
Assess potential superiority of this regimen versus historical controls with melphalan and prednisone alone | 2 years
Evaluate efficacy in terms of progression-free survival and overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: San Miguel Jesús, Professor, Study Chair — Hospital Clinico Universitario de Salamanca
Locations (19):
- Spain (19):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - Hospital Doce de Octubre, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Morales Messeguer, Murcia, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínic, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Virgen Blanca de León, León
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital General de Segovia, Segovia

REFERENCES:
- [Background] Greenlee RT, Murray T, Bolden S, Wingo PA. Cancer statistics, 2000. CA Cancer J Clin. 2000 Jan-Feb;50(1):7-33. doi: 10.3322/canjclin.50.1.7. PMID 10735013
- [Background] 2. Longo D. Plasma cell disorders. In : Fauce A, et al. Ed. Harrison's Principles of Internal Medicine. 14th Ed. New York, New York: Mc Graw-Hill; 1998: 712-718
- [Background] Raje N, Anderson K. Thalidomide--a revival story. N Engl J Med. 1999 Nov 18;341(21):1606-9. doi: 10.1056/NEJM199911183412110. No abstract available. PMID 10564693
- [Background] Oken MM. Management of Myeloma: Current and Future Approaches. Cancer Control. 1998 May;5(3):218-225. doi: 10.1177/107327489800500302. PMID 10761055
- [Background] Westin J. Conventional chemotherapy in multiple myeloma. Pathol Biol (Paris). 1999 Feb;47(2):169-71. PMID 10192883
- [Background] Huang YW, Hamilton A, Arnuk OJ, Chaftari P, Chemaly R. Current drug therapy for multiple myeloma. Drugs. 1999 Apr;57(4):485-506. doi: 10.2165/00003495-199957040-00004. PMID 10235689
- [Background] Smith ML, Newland AC. Treatment of myeloma. QJM. 1999 Jan;92(1):11-4. doi: 10.1093/qjmed/92.1.11. PMID 10209667
- [Background] Bataille R, Harousseau JL. Multiple myeloma. N Engl J Med. 1997 Jun 5;336(23):1657-64. doi: 10.1056/NEJM199706053362307. No abstract available. PMID 9171069
- [Background] Alexanian R, Dimopoulos M. The treatment of multiple myeloma. N Engl J Med. 1994 Feb 17;330(7):484-9. doi: 10.1056/NEJM199402173300709. No abstract available. PMID 8289856
- [Background] Gregory WM, Richards MA, Malpas JS. Combination chemotherapy versus melphalan and prednisolone in the treatment of multiple myeloma: an overview of published trials. J Clin Oncol. 1992 Feb;10(2):334-42. doi: 10.1200/JCO.1992.10.2.334. PMID 1531068
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Alexanian R, Dimopoulos MA, Delasalle K, Barlogie B. Primary dexamethasone treatment of multiple myeloma. Blood. 1992 Aug 15;80(4):887-90. PMID 1498331
- [Background] Case DC Jr, Lee DJ 3rd, Clarkson BD. Improved survival times in multiple myeloma treated with melphalan, prednisone, cyclophosphamide, vincristine and BCNU: M-2 protocol. Am J Med. 1977 Dec;63(6):897-903. doi: 10.1016/0002-9343(77)90543-5. No abstract available. PMID 605911
- [Background] Attal M, Harousseau JL, Stoppa AM, Sotto JJ, Fuzibet JG, Rossi JF, Casassus P, Maisonneuve H, Facon T, Ifrah N, Payen C, Bataille R. A prospective, randomized trial of autologous bone marrow transplantation and chemotherapy in multiple myeloma. Intergroupe Francais du Myelome. N Engl J Med. 1996 Jul 11;335(2):91-7. doi: 10.1056/NEJM199607113350204. PMID 8649495
- [Background] Driscoll J. The role of the proteasome in cellular protein degradation. Histol Histopathol. 1994 Jan;9(1):197-202. PMID 8003815
- [Background] Richter-Ruoff B, Wolf DH. Proteasome and cell cycle. Evidence for a regulatory role of the protease on mitotic cyclins in yeast. FEBS Lett. 1993 Dec 20;336(1):34-6. doi: 10.1016/0014-5793(93)81603-w. PMID 8262212
- [Background] Goldberg AL, Stein R, Adams J. New insights into proteasome function: from archaebacteria to drug development. Chem Biol. 1995 Aug;2(8):503-8. doi: 10.1016/1074-5521(95)90182-5. PMID 9383453
- [Background] Hideshima T, Richardson P, Chauhan D, Palombella VJ, Elliott PJ, Adams J, Anderson KC. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001 Apr 1;61(7):3071-6. PMID 11306489
- [Background] Sherr CJ. Cancer cell cycles. Science. 1996 Dec 6;274(5293):1672-7. doi: 10.1126/science.274.5293.1672. PMID 8939849
- [Background] Koepp DM, Harper JW, Elledge SJ. How the cyclin became a cyclin: regulated proteolysis in the cell cycle. Cell. 1999 May 14;97(4):431-4. doi: 10.1016/s0092-8674(00)80753-9. No abstract available. PMID 10338207
- [Background] Read MA, Neish AS, Luscinskas FW, Palombella VJ, Maniatis T, Collins T. The proteasome pathway is required for cytokine-induced endothelial-leukocyte adhesion molecule expression. Immunity. 1995 May;2(5):493-506. doi: 10.1016/1074-7613(95)90030-6. PMID 7538441
- [Background] Palombella VJ, Rando OJ, Goldberg AL, Maniatis T. The ubiquitin-proteasome pathway is required for processing the NF-kappa B1 precursor protein and the activation of NF-kappa B. Cell. 1994 Sep 9;78(5):773-85. doi: 10.1016/s0092-8674(94)90482-0. PMID 8087845
- [Background] Zetter BR. Adhesion molecules in tumor metastasis. Semin Cancer Biol. 1993 Aug;4(4):219-29. PMID 8400144
- [Background] Beg AA, Baltimore D. An essential role for NF-kappaB in preventing TNF-alpha-induced cell death. Science. 1996 Nov 1;274(5288):782-4. doi: 10.1126/science.274.5288.782. PMID 8864118
- [Background] Baldwin AS. Control of oncogenesis and cancer therapy resistance by the transcription factor NF-kappaB. J Clin Invest. 2001 Feb;107(3):241-6. doi: 10.1172/JCI11991. No abstract available. PMID 11160144
- [Background] 26. McConkey DJ, Pettaway C, Elliott P, et al. The proteasome as a new drug target in metastatic prostate cancer. ATMDACC 7th Annual Genitourinary Oncology Conference, 1998
- [Background] Adams J, Palombella VJ, Sausville EA, Johnson J, Destree A, Lazarus DD, Maas J, Pien CS, Prakash S, Elliott PJ. Proteasome inhibitors: a novel class of potent and effective antitumor agents. Cancer Res. 1999 Jun 1;59(11):2615-22. PMID 10363983
- [Background] 28. Millenium Pharmaceuticals, Inc. (PS-341) Investigator's Brochure, Version 5.0, 2001
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Mileshkin L, Biagi JJ, Mitchell P, Underhill C, Grigg A, Bell R, McKendrick J, Briggs P, Seymour JF, Lillie K, Smith JG, Zeldis JB, Prince HM. Multicenter phase 2 trial of thalidomide in relapsed/refractory multiple myeloma: adverse prognostic impact of advanced age. Blood. 2003 Jul 1;102(1):69-77. doi: 10.1182/blood-2002-09-2846. Epub 2003 Mar 13. PMID 12637329
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Blade J, Samson D, Reece D, Apperley J, Bjorkstrand B, Gahrton G, Gertz M, Giralt S, Jagannath S, Vesole D. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. Myeloma Subcommittee of the EBMT. European Group for Blood and Marrow Transplant. Br J Haematol. 1998 Sep;102(5):1115-23. doi: 10.1046/j.1365-2141.1998.00930.x. No abstract available. PMID 9753033
- See also: Spanish association of Haematology — http://www.aehh.org